CLINICAL TRIAL: NCT06439108
Title: Single Versus Double Symphyseal Plating in Management of Vertically Unstable Open Book Pelvic Ring Injuries: A Randomized Controlled Trial
Brief Title: Single vs Double Symphyseal Plating in Management of Vertically Unstable Open Book Pelvic Ring Injuries:
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Islam Moussa, lecturer of orthopedic surgery, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R65/2023
Record Dates: First submitted 2024-05-26; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Evaluation of Single Symphyseal Plating in APC III Injuries
Keywords: APC III pelvic ring injuries; single symphyseal plating; double symphyseal plating; functional outcome; Majeed pelvic score

STUDY DESIGN:
Intervention Model Description: An independent doctor created the randomization sequence using Excel 2016 (computerized random numbers) with a 1:1 allocation via random block sizes of 2, 4, and 6; he assigned the sample numbers equally to each group and assigned the block. Patients and physicians allocated to each intervention group were aware of the allocation; however, the data analysts and the outcome assessors were kept blinded to the allocation. The investigators prospectively carried out this study on 30 patients with APC III pelvic ring injuries between March 2022 and May 2023 that met our inclusion criteria. The independent doctor allocated the 30 cases to two groups: Group A (15 cases): single superior symphyseal plate, group B (15 cases): double superior & anterior symphyseal plate
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients and physicians allocated to each intervention group were aware of the allocation; however, the data analysts and the outcome assessors were kept blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single superior symphyseal plate (Active Comparator): 15 cases undergoing single superior symphyseal plate, reduction of the posterior ring was either closed reduction in SI joint dislocations & fracture-dislocations and sacral fractures or open reduction in iliac wing fractures through the lateral window of the ilioinguinal approach.Anterior pelvic ring reduction and fixation was done via the classic Pfannenstiel approach
  Interventions: Procedure: single symphyseal plating in management of vertically unsable open book pelvic ring injuries
- double superior & anterior symphyseal plates (Active Comparator): 15 cases undergoing double superior & anterior symphyseal plates, 15 cases undergoing double superior & anterior symphyseal plates, reduction of the posterior ring was either closed reduction in SI joint dislocations & fracture-dislocations and sacral fractures or open reduction in iliac wing fractures through the lateral window of the ilioinguinal approach.Anterior pelvic ring reduction and fixation was done via the classic Pfannenstiel approach
  Interventions: Procedure: single symphyseal plating in management of vertically unsable open book pelvic ring injuries

INTERVENTIONS:
Procedure: single symphyseal plating in management of vertically unsable open book pelvic ring injuries — open book pelvic ring injuries can be managed via the two techniques.
  Other Names: double symphyseal plating in management of vertically unsable open book pelvic ring injuries

SUMMARY:
compare functional, radiological outcomes, implant failure and the incidence of recurrent diastasis of single superior symphyseal plate versus double plating in management of vertically unstable open book injuries

DETAILED DESCRIPTION:
The real algorithm was the necessity for double superior & anterior plating versus single superior symphyseal plate in management of APC III pelvic ring injuries, whether the incidence of intraoperative and short-term postoperative complications, recurrent diastasis, radiological and functional outcomes differed between these two methods. Our hypothesis was that the use of an additional anterior symphyseal plating could provide a more rigid fixation, with less complications of recurrent diastasis or implant failure. Also it will be applied through the same incision without increasing the patient overall morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Anterior ring symphyses diastasis
* Tile C pelvic ring injuries
* Age between 16-60 years' old

Exclusion Criteria:

* Tile B pelvic ring injuries
* Isolated bony fractures of the anterior pelvic ring
* Open fractures
* Age less than 14 years and older than 60 years
* Associated internal organ injuries that require definitive intervention

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Rate of Excellent, Good, Fair or Poor clinical outcome | 1 year postoperative
  clinical assessment by Majeed pelvic scoring system evaluated and calculated at each follow-up visit with the mean value presented
Rate of Excellent, Good, Fair or Poor radiological outcome | 1 year postoperative
  Radiological assessment using Matta & Tornetta radiological principles via plain x-ray pelvis showing both hips: anteroposterior, inlet and outlet views & CT pelvis if available; we evaluated five criteria on X-ray films postoperatively: residual posterior displacement, vertical displacement, pubic symphyseal translation, sagittal rotation, and gapping of the sacroiliac joint; according to the grading of Matta and Tornetta, we classified the results into Excellent (less than or equal 4 mm), Good (4-10 mm), Fair (10-20 mm), and Poor (more than 20 mm).
Rate of recurrent diastasis | throughout study completion, average one year postoperative
  rate of symphyseal translation was measured & compared between the two study groups

SECONDARY OUTCOMES:
Mean intraoperative blood loss | up to 5 days post-operative
  The mean blood loss was calculated in milliliters and compared between the two study groups, it was measured intraoperative and postoperative from suction drains
Mean operative time | It was calculated intra-operative
  The mean operation time was calculated in minutes and compared between the two study groups
postoperative complications' rate | 1 year post-operative
  We focused the evaluation of Postoperative complications on the local complications related to fixation principles and technique: LLD, implant failure, wound infection, residual malunion or non-union of the anterior ring, and loss of reduction (2ry SI dislocation or any rotational or vertical re-displacement)

CONTACTS AND LOCATIONS:
Overall Officials: Islam S Moussa, MD, Study Chair — no funding recieved
Locations (1):
- Islam Sayed Moussa, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
share the plan
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: full access

REFERENCES:
- [Derived] Moussa IS, Abdelmonem IM, Nagy AM. Single versus double symphyseal plating in management of tile C1-2 and C1-3 pelvic ring injuries: a randomized controlled trial. BMC Surg. 2025 May 9;25(1):200. doi: 10.1186/s12893-025-02936-3. PMID 40346505